CLINICAL TRIAL: NCT01789931
Title: Examination of a New Non Invasive Sensor "Lifebeam" During HTT (Heat Tolerance Test) in Protective Clothing
Brief Title: Examination of a New Non Invasive Sensor "Lifebeam" During HTT in Protective Clothing
Acronym: lifebeam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Barliz Adato, head investigator of Heller institute of physiology, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-12-9435-BA-CTIL
Record Dates: First submitted 2012-12-06; First posted 2013-02-12 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Heat Illness
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Research arm (Experimental): The participants will undergo an examination day in which they will complete VO2max test to evaluate their aerobic fitness. Afterwards they'll undergo 3 heat tolerance test (HTT) days: without CB protective clothing, with CB protective clothing, and with work clothes. During the tests, a "Lifebeam" sensor will be attached to their skin.
  Interventions: Device: "Lifebeam"

INTERVENTIONS:
Device: "Lifebeam" — The "lifebeam" sensor will be attached to the participant's skin during the HTT.

SUMMARY:
CB (Chemical Biological)protective clothing provides a thermal resistance between the human body and its environment. CB protective clothing will be essential for combat soldiers in case of non conventional attacks. "Lifebeam" developed a new non invasive sensor for body core temperature detection. The research purpose is to evaluate the "Lifebeam" sensor during heat tolerance test while wearing CB protective clothing.

ELIGIBILITY:
Inclusion Criteria:

* age 21-30
* healthy
* after medical checkup
* after signing concent form

Exclusion Criteria:

* heart disease
* respiratory disease
* baseline bp above 140/90 mmHg
* sleep disorders
* diabetes
* anhydrosis
* skin disease
* acute illness in last 3 days prior to the examination

Ages: 21 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Heat tolerance test | 1 year
  The test is performed in a climatic chamber at a temperature of 40oC and 40% relative humidity. During the test, the subject walks on a treadmill at a speed of 5 km/hr at a 2% grade for 2h. Body core temperature and heart rate are continuously monitored, and sweat rate is computed from body weight prior to and after the test, corrected for fluid intake. Heat intolerance is determined when body core temperature elevates above 38.5oC, when heart rate elevates above 150 bpm, or when either does not tend to reach a plateau.
VO2 test | 1 year
  Volunteer's oxygen consumption (VO2) will be monitored continuously with a metabolic chart (ZAN), while running for 10 min on a treadmill under comfortable environmental conditions.

SECONDARY OUTCOMES:
Skin temperature | 1 year
  The volunteers will undergo heat tolerance test. Their skin temperature will be measured by skin thermistors and will be monitored continuously and viewed by the attending medical staff. Automatically all data will be recorded by the monitoring Biopac system.
Rectal temperature | 1 year
  The volunteers will undergo heat tolerance test. Their rectal temperature will be measured by rectal thermistor and will be monitored continuously and viewed by the attending medical staff. Automatically all data will be recorded by the monitoring Biopac system.
Heart rate | 1 year
  During the HTT and the VO2 test heart rates will be monitored continuously and will be stored by a heart rate wristwatch, (POLAR, Finland).
blood circulation parameters | 1 year
  Evaluation by the optic sensor "Lifebeam" of the blood circulation parameters (heart rate, blood flow velocity, perfusion, and ventilation rate) in the peripheral arterioles

CONTACTS AND LOCATIONS:
Overall Officials: Barliz Adato, MD, Principal Investigator — Heller institute, Sheba medical center
Locations (1):
- Sheba medical center, Tel-Hashomer, Ramat- Gan, Israel